CLINICAL TRIAL: NCT04490811
Title: Seroprevalence and Immunoprotection Against SARS-CoV2 in Children Hospitalized in Paris
Brief Title: Seroprevalence and Immunoprotection Against COVID-19 in Parisian Children
Acronym: AP-PEDCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Principal Investigator, Isabelle Sermet-Gaudelus, Professor, Hôpital Necker-Enfants Malades
Other Study IDs: HNeckerNM
Record Dates: First submitted 2020-06-20; First posted 2020-07-29 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention. observational cohort study — blood sampling is part of care
  Other Names: no intervention

SUMMARY:
The paediatric population present mild or asymptomatic form of SARS-CoV-2 infection. This study asses the frequency of patients with SARS-CoV2 Antibodies (Ab) (seroprevalence) and the neutralizing typology of those Ab (immunoprotection) in children from 7 days to 18 years of age hospitalized for no more than 4 days and whose clinical status requires blood sample regardless of the symptoms Patients are included on a given day, after information, before blood sampling performed as part of the care. 500 µL of sera, normally discarded will be kept to perform SARS-Cov2 serology.

DETAILED DESCRIPTION:
Background of the study:

The fraction of undiagnosed cases is a critical epidemiological characteristic that modulates the epidemic potential of SARS-CoV-2 emerging respiratory virus. These subjects most often present themselves in benign or totally asymptomatic form, although they are likely to spread the virus in the general population. The containment strategy was implemented in France to reverse the exponential epidemic growth of infection.

A crucial issue is the specific study of the paediatric population because the prevalence of symptomatic infections is low and children are mostly mild and under-diagnosed. Children could frequently be asymptomatic carriers and act as a real reservoir for the spread of the virus. In these "sub-symptomatic" carriers, the viral load may be low, and it is possible that PCR nasal tests may be defective. The serological study is therefore essential because it will inform us about the speed and effectiveness of seroconversion and therefore about the immunoprotection of this subpopulation.

The rationale for the study is that the proportion of children who have developed immunoprotection is decisive in defining measures to control the epidemic. It is essential to assess the prevalence and typology of antibody responses in this population and to follow kinetics over time.

The many emerging atypical forms and in particular the post-infectious kawasaki-like forms have a very particular immunopathological profile that provides information on the natural history of the disease.

Main objectives of the study to assess the prevalence of seroconversion (seroprevalence) in a pediatric population sample to study the immunopathological profile of clinical forms attributed to SARS-CoV-2 infection

Design of the study Patients are included on a given day, after information, before blood sampling performed as part of the care. 500 µL of sera, normally discarded will be kept to perform SARS-Cov2 serology. According to data currently collected in France, 5% of children taken from symptoms are infected. Given that nasopharyngeal testing is lacking in this pediatric population, we anticipate an increase in the number of subjects who have been infected or have an ongoing infection at least 10%. A sample of 800 subjects will therefore include at least 80 children with infection.

A questionnaire will extract relevant variables to this project:

* Any symptoms of the index case or his family since December 2019 consistent with COVID-19
* Comorbidities and treatment
* Reason for hospitalization
* History of contact case
* Clinical signs on the day of collection
* Result of RT-PCT SARS-CoV2 nasopharyngeal if made in the index case

ELIGIBILITY:
Inclusion Criteria:

* any child over 7 days and under 18 years of age who has been hospitalized for no more than 4 days and who has a blood sample regardless of the symptoms;

Exclusion Criteria:

* Any child under 7 days

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All hospitalized children at Assistance Publique Hôpitaux de Paris
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
serological test | 48 weeks
  Ab against SARS-CoV-2

SECONDARY OUTCOMES:
neutralizing Ab | 48 weeks
  activity of the antibodies against SARS-CoV2
Immuno phenotyping | 48 weeks
  Lymphocyte response phenotyping

CONTACTS AND LOCATIONS:
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No